CLINICAL TRIAL: NCT07115056
Title: Extended Post-Operative Oral Tranexamic Acid Dosing After ACL Reconstruction: A Multicenter Randomized Controlled Trial
Brief Title: Extended Oral Tranexamic Acid After Anterior Cruciate Ligament Reconstruction
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Campbell Clinic (Other)
Collaborators: Duke University (Other); University of Pittsburgh (Other); Endeavor Health (Other); University of Cincinnati (Other); Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Frederick Azar, Chief of Staff, Campbell Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Oral TXA After ACL-R
Record Dates: First submitted 2025-07-30; First posted 2025-08-11 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: ACL Injury; ACL Tears; ACL Surgery
Keywords: ACL; ACL Repair; ACL Reconstruction; TXA; tranexamic acid
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral TXA (Experimental): Participants in this arm will receive oral tranexamic acid (TXA), 1.95 g daily (three 650 mg capsules) from POD 1 to POD 10, for a total of 10 doses (30 capsules). All participants will also receive 1 g IV TXA before incision and 1 g IV TXA at surgical closure as part of standard care.
  Interventions: Drug: Tranexamic Acid (TXA)
- Placebo (Placebo Comparator): Participants in this arm will receive oral placebo capsules (microcrystalline cellulose), 3 capsules daily from postoperative day (POD) 1 to POD 10, for a total of 10 doses (30 capsules). All participants will also receive 1 g IV TXA before incision and 1 g IV TXA at surgical closure as part of standard care.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) — Oral tranexamic acid (TXA) is administered at a dose of 1.95 grams per day, divided into three 650 mg capsules taken once daily, starting on postoperative day (POD) 1 through POD 10 (10 total doses; 30 capsules) to the treatment group.
  Arms: Oral TXA
Drug: Placebo — Participants in this arm will receive oral placebo capsules (microcrystalline cellulose), 3 capsules daily from postoperative day (POD) 1 to POD 10, for a total of 10 doses (30 capsules).
  Arms: Placebo

SUMMARY:
This is a prospective, multi-center, randomized, double-blind, placebo-controlled trial evaluating the efficacy of oral tranexamic acid (TXA) in improving postoperative outcomes following anterior cruciate ligament reconstruction (ACLR) using patellar tendon autograft in adolescent and young adult patients.

A total of 100 patients, aged 14 to 22 years and undergoing eligible ACLR, will be enrolled across multiple participating sites. Eligible participants will be randomized 1:1 to receive either oral TXA (1.95 g per day, divided into three 650 mg capsules) or placebo (microcrystalline cellulose) once daily from postoperative day 1 to 10, in addition to standard intraoperative care. All participants will receive 1 g IV TXA prior to incision and 1 g IV TXA at closure, per standard surgical protocol.

The primary outcome is improvement in postoperative pain, as measured by the Visual Analog Scale (VAS). Secondary outcomes are knee range of motion, quadriceps strength, isokinetic strength, time to straight leg raise, time to return to sport, International Knee Documentation Committee score, Lyshom score, and morphine milligram equivalents. Participants will be followed through routine postoperative visits at the participating institutions out to one year with a phone call for patient reported outcomes at 2 years.

DETAILED DESCRIPTION:
This multi-center, prospective, randomized, double-blind, placebo-controlled clinical trial is designed to evaluate the effect of oral tranexamic acid (TXA) on postoperative outcomes following anterior cruciate ligament reconstruction (ACLR) using bone-tendon-bone (BTB) autograft in adolescent and young adult patients.

Background:

Tranexamic acid is a synthetic antifibrinolytic agent that competitively inhibits plasminogen activation, helping to reduce bleeding. IV TXA is routinely used during orthopedic procedures, including ACLR, and has been shown to reduce intraoperative blood loss. However, the benefit of extending antifibrinolytic coverage with oral TXA in the early postoperative period has not been well studied in this population. This trial aims to investigate whether a 10-day postoperative course of oral TXA improves pain and recovery outcomes following ACLR.

Study Design:

Participants will be randomized in a 1:1 ratio to receive either oral TXA or a placebo. Randomization will be conducted using computer-generated allocation. Both the participants and the study team will remain blinded to group assignment.

Group A (Placebo): Participants will receive 10 doses (30 capsules total) of microcrystalline cellulose (placebo), to be taken daily from postoperative day (POD) 1 through POD 10.

Group B (Oral TXA): Participants will receive 10 doses (30 capsules total) of oral TXA, dosed at 1.95 g per day (650 mg per capsule, 3 capsules daily) from POD 1 through POD 10.

All participants will receive standard intraoperative care, including 1 gram IV TXA prior to skin incision and an additional 1 gram IV TXA at surgical closure. Postoperative pain management will be administered per standard clinical practice and at the discretion of the treating surgical team.

Patient Population:

The study will enroll 100 patients aged 14 to 22 years undergoing isolated ACLR with a BTB autograft at Campbell Clinic Surgery Center and collaborating study sites.

Study Procedures:

Eligible patients will be identified via chart review and approached in clinic or via phone. Informed consent (and assent where applicable) will be obtained during a routine preoperative visit. Baseline data will be collected, including demographics and medical history. Participants will then be randomized and provided with study medication (oral TXA or placebo) to begin on POD 1.

Outcomes: The primary outcome is improvement in postoperative pain, as measured by the Visual Analog Scale (VAS). Secondary outcomes are knee range of motion, quadriceps strength, isokinetic strength, time to straight leg raise, time to return to sport, International Knee Documentation Committee score, Lyshom score, and morphine milligram equivalents.

Blinding and Allocation:

All capsules will be identical in appearance and packaging to maintain blinding. Randomization will be performed centrally and allocation concealed. Study staff, treating physicians, and patients will remain blinded until data analysis.

Safety Monitoring:

Participants will be monitored for adverse events throughout the study period. TXA is generally well tolerated but may pose thrombotic risk in susceptible individuals; exclusion criteria are designed to minimize this risk. The study team will report any serious adverse events (SAEs) to the IRB per institutional guidelines.

The study is powered to detect clinically meaningful differences in VAS scores, with a planned enrollment of 50 patients per group, allowing for a 20% loss to follow-up. This trial aims to clarify the role of extended postoperative oral TXA in reducing inflammation, pain, and bleeding in young ACLR patients, potentially offering a low-cost adjunct to current perioperative care.

ELIGIBILITY:
Inclusion Criteria:

* 14-22 year old individuals with ACL tear undergoing primary ACLR with patellar tendon autograft.
* Closed or closing proximal tibial and distal femoral physes on pre-operative radiographs (less than one year of growth remaining based on MRI and radiographic bone age assessment)
* Fluent in English
* Willing to participate
* Patient weight greater than or equal to 100lbs (45.4kg)

Exclusion Criteria:

* Revision ACLR, multi-ligamentous knee reconstruction, inclusion of lateral extra-articular tenodesis (LET) or Anterolateral Ligament (ALL) reconstruction
* Concomitant meniscal repair or chondral preservation surgery requiring postoperative limited weightbearing status (nonweightbearing or partial weightbearing)
* Have a prior history of deep vein thrombosis (DVT) or thromboembolic event
* Known allergy or hypersensitivity to TXA
* Using combination hormonal contraception

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Pre-op and 2 week, 6 week, 12 week, 6 months, 1 year, 2 year post op
  The Visual Analog Scale (VAS) is a validated patient-reported outcome measure used to assess pain intensity. Patients rate their pain on a scale from 0 (no pain) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Knee Range of Motion | Pre-op and 2-week, 6-week, 12-week, 6 months, 1-year post-op
  Knee range of motion (ROM) will be assessed during visits using a goniometer to measure flexion and extension.
Quadriceps Strength | Pre-op and 2-week, 6-week, 12-week, 6 months, 1-year post-op
  Quadriceps strength will be assessed using a dynamometer.
Isokinetic Strength | 6 months, 9 months, 1-year post-op
  Isokinetic strength will be tested through biodex testing.
Time to Straight Leg Raise | Up to 1 year
  Time to Straight Leg Raise (SLR) is defined as the number of days from surgery to the first postoperative day on which the patient can perform an active straight leg raise without an extensor lag.
Time to Return to Sport | Up to 1 year
  Time to Return to Sport is defined as the number of days from surgery to the patient's clearance to resume full participation in sport-specific activities. Clearance is determined by the treating provider based on clinical evaluation, functional testing, and rehabilitation progress. This measure reflects overall recovery and readiness to return to pre-injury activity levels.
International Knee Documentation Committee Score | Pre-op and 6 months, 1-year, 2-years post-op
  The International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form is a validated, patient-reported outcome measure used to assess symptoms, function, and sports activity in individuals with knee disorders. Scores range from 0 to 100, with higher scores indicating better function and fewer symptoms.
Lysholm Knee Score | Pre-op and 6 months, 1-year, 2-years post-op
  The Lysholm Knee Scoring Scale is a validated, patient-reported outcome measure used to assess knee function, symptoms, and stability following ligament injuries. Scores range from 0 to 100, with higher scores indicating better knee function.
Morphine Milligram Equivilants | 2 weeks following surgery
  Morphine Milligram Equivalents (MMEs) will be used to quantify opioid consumption in the postoperative period (2 weeks post-op). All prescribed and consumed opioid medications will be converted to MMEs using standard CDC conversion factors. Total MMEs will be calculated for each participant over the initial postoperative period.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Endeavor Health, Evanston, Illinois
  - Washington University School of Medicine in St. Louis, Chesterfield, Missouri
  - Duke University School of Medicine, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Campbell Clinic, Germantown, Tennessee

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to concerns about participant privacy and confidentiality, limitations in resources to properly de-identify and manage data sharing, and institutional policies restricting data access. These measures are in place to ensure compliance with ethical standards and protect sensitive participant information.

REFERENCES:
- [Background] Vermeijden HD, Yang XA, Rademakers MV, Kerkhoffs GMMJ, van der List JP, DiFelice GS. Early and Delayed Surgery for Isolated ACL and Multiligamentous Knee Injuries Have Equivalent Results: A Systematic Review and Meta-analysis. Am J Sports Med. 2023 Mar;51(4):1106-1116. doi: 10.1177/03635465211069356. Epub 2022 Jan 31. PMID 35099334
- [Background] Tan TK, Ng KT, Lim HJ, Radic R. Effect of tranexamic acid in arthroscopic anterior cruciate ligament repair: A systematic review and meta-analysis of randomised clinical trials. J Orthop Surg (Hong Kong). 2021 May-Aug;29(2):23094990211017352. doi: 10.1177/23094990211017352. PMID 34027721
- [Background] Romereim SM, Smykowski MR, Ball EK, Carey EG, Cuadra M, Williams A, Hickson K, Haim K, Sumith M, Yu Z, Jin G, Foureau D, Steuerwald N, Odum S, Fearing BV, Riboh JC. Immunophenotyping of Synovial Tissue in Adolescents Undergoing ACL Reconstruction: What Is the Role of Synovial Inflammation in Arthrofibrosis? Am J Sports Med. 2025 Feb;53(2):315-326. doi: 10.1177/03635465241305411. Epub 2025 Jan 7. PMID 39772756
- [Background] Kirwan MJ, Diltz ZR, Dixon DT, Rivera-Peraza CA, Gammage CJ, Mihalko WM, Harkess JW, Guyton JL, Crockarell JR, Ford MC. The AAHKS Clinical Research Award: Extended Postoperative Oral Tranexamic Acid in Total Knee Arthroplasty: A Randomized Controlled Pilot Study. J Arthroplasty. 2024 Sep;39(9S2):S13-S17. doi: 10.1016/j.arth.2024.02.073. Epub 2024 Feb 29. PMID 38430972
- [Background] Keays SL, Mellifont DB, Keays AC, Stuelcken MC, Lovell DI, Sayers MGL. Long-term Return to Sports After Anterior Cruciate Ligament Injury: Reconstruction vs No Reconstruction-A Comparison of 2 Case Series. Am J Sports Med. 2022 Mar;50(4):912-921. doi: 10.1177/03635465211073152. Epub 2022 Feb 11. PMID 35148249
- [Background] Goldstein K, Jones C, Kay J, Shin J, de Sa D. Tranexamic Acid Administration in Arthroscopic Surgery Is a Safe Adjunct to Decrease Postoperative Pain and Swelling: A Systematic Review and Meta-analysis. Arthroscopy. 2022 Apr;38(4):1366-1377.e9. doi: 10.1016/j.arthro.2021.10.001. Epub 2021 Oct 14. PMID 34655767
- [Background] Felli L, Revello S, Burastero G, Gatto P, Carletti A, Formica M, Alessio-Mazzola M. Single Intravenous Administration of Tranexamic Acid in Anterior Cruciate Ligament Reconstruction to Reduce Postoperative Hemarthrosis and Increase Functional Outcomes in the Early Phase of Postoperative Rehabilitation: A Randomized Controlled Trial. Arthroscopy. 2019 Jan;35(1):149-157. doi: 10.1016/j.arthro.2018.07.050. PMID 30611343
- [Background] Cen L, Liu H, Li M, Zhang YF, Zhang HJ, Huang ZY. Intraoperative tranexamic acid reduces postoperative haemarthrosis and improves early functional outcomes in double-bundle anterior cruciate ligament reconstruction. J Orthop. 2024 Dec 10;65:51-56. doi: 10.1016/j.jor.2024.12.005. eCollection 2025 Jul. PMID 39801905